CLINICAL TRIAL: NCT01261715
Title: Staples Versus Dermabond for Closure of the Skin After Cesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Meir Medical Center (Other)
Responsible Party: Sadeh Dana MD, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 155-2010
Record Dates: First submitted 2010-12-06; First posted 2010-12-16 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-10

CONDITIONS: Cesarean Section Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Woman with previous ceasarean section - staples (Active Comparator)
  Interventions: Procedure: Dermabond- liquid skin adhesive

INTERVENTIONS:
Procedure: Dermabond- liquid skin adhesive — Dermabond- liquid skin adhesive

SUMMARY:
Two of the more frequently used options for skin closure following a cesarean delivery include staples or sutures (stitches). Another method of closure is Dermabond- liquid skin adhesive. This method of closure is used less frequently than either staples or sutures.

Few studies have been done regarding whether Dermabond is preferable or affect the outcome of a cesarean section surgery. The aim of our study is to find weather Dermabond haas better result for the closure of cesarean section wounds.

ELIGIBILITY:
Inclusion Criteria:

Woman over 18 year Woman having elective caesarean section

Exclusion Criteria:

Age under 18 Woman having an emergency caesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Cosmetic objective evaluation of the scar | 6 weeks postoperatively

SECONDARY OUTCOMES:
The difference in pain between the two type of closure | 1 and 4 days postoperatively
The difference in patient satisfaction with the scar result | 6 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Dana Sadeh, MD, Principal Investigator — MD
Locations (1):
- Meir medical center, Kfar Saba, Israel